CLINICAL TRIAL: NCT06054997
Title: Anaesthesiologic Considerations for Intraoperative ECMO Anticoagulation During Lung Transplantation: A Single-centre, Retrospective, Observational Study
Brief Title: Anaesthesiologic Considerations for Intraoperative ECMO Anticoagulation During Lung Transplantation
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Jaromir Vajter, Head of ECLS Center, Principal Investigator, University Hospital, Motol
Other Study IDs: LUTX-UFH
Record Dates: First submitted 2023-09-07; First posted 2023-09-26 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Lung Transplantation
Keywords: ECMO; Lung transplantation; heparin; UFH; ROTEM; anticoagulation; anesthesiology; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lower dose UFH/kg group: UFH below or equal to 60 IU/kg/surgery
- higher dose UFH/kg group: UFH above 60 IU/kg/surgery

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a frequently used extracorporeal support measure during the intraoperative period in lung transplantation. A certain amount of anticoagulation, mainly unfractionated heparin (UFH), is used as part of ECMO support. One of the most common perioperative complications during lung transplantation is bleeding. An inadequately high dose of UFH can increase the risk of bleeding. In this study, the investigators hypothesised that a lower dose of UFH would decrease the risk of nonsurgical bleeding complications during lung transplantation and would not pose an increased risk of thrombotic complications for patients or ECMO circuits.

DETAILED DESCRIPTION:
This study was designed as a single-centre, retrospective, observational study including all lung transplants between January 2020 and December 2022 within the Prague Lung Transplant Program Motol University Hospital. A total of 141 patients were transplanted during the study period. The exclusion criteria were lung transplant without intraoperative ECMO support, block heart-lung transplantation, ECMO bridge to lung transplant and planned postoperative ECMO. The inclusion criteria were lung transplantation performed with intraoperative ECMO support, central ECMO cannulation, and successful ECMO support termination at the end of the surgery. According to the study inclusion criteria, only lung transplants under intraoperative central ECMO cannulation with successful ECMO weaning were included. A total of 109 patients fulfilled the inclusion criteria. Thirty-two patients were excluded based on the following exclusion criteria: heart-lung transplant (HLTx) n=4, ECMO bridge n=4, transplantation (Tx) without ECMO n=8, and planned prolonged ECMO n=16. UFH was used for ECMO anticoagulation in all patients. The subjects were divided into two groups according to the UFH dose during the entire surgical procedure. In the first group, the dose of UFH was below or equal to 60 IU/kg/surgery. In the second group, the dose of UFH was above 60 IU/kg/surgery. A cut-off value of 60 IU/kg was determined according to the available literature review. Values ≤ 60 IU/kg/surgery were considered relatively lower doses, and values > 60 IU/kg/surgery were considered higher doses of UFH. The UFH effect was monitored by activated clotting time (ACT) values. The intraoperative haemoglobin level target for red blood cells (RBCs) substitution was 100 g/l. The parameters that will be monitored intraoperatively in both groups are the total blood loss in millilitres and related to the patient's weight during the operation, the total amount of UFH administered to the patient during the procedure in international units (IU) and related to the patient's weight, and the consumption of blood derivatives during surgery such as red blood cells, fresh frozen plasma (FFP) and platelets. In both groups, ACT values will be monitored after the administration of UFH before ECMO cannulation. In the postoperative period, the investigators will monitor the development of hemothorax requiring surgical revision. The investigators consider surgical revision for hemothorax to be a significant bleeding complication. 30-day and 90-day mortality, ECMO- and patient-related thrombotic complications will be assessed.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria were lung transplantation performed with intraoperative ECMO support, central ECMO cannulation, and successful ECMO support termination at the end of the surgery.

Exclusion Criteria:

- The exclusion criteria were lung transplant without intraoperative ECMO support, block heart-lung transplantation, ECMO bridge to lung transplant and planned postoperative ECMO.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All lung transplants between January 2020 and December 2022 within the Prague Lung Transplant Program Motol University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Outcome Measure intraoperative blood loss | intraoperative
  Change in the amount of intraoperative blood loss (from the start of the surgical procedure till the end of the procedure)

SECONDARY OUTCOMES:
Outcome Measure the consumption of blood derivatives | intraoperative
  Change in the intraoperative blood derivatives consumption (from the start of the surgical procedure till the end of the procedure)
Outcome Measure surgical revision for postoperative bleeding | From enrollment to 90-day
  Change in frequency of the surgical revision for postoperative bleeding (From enrollment to 90-day)
Outcome Measure thrombotic complications | intraoperative
  Change in frequency of the intraoperative thrombotic complications (from the start of the surgical procedure till the end of the procedure)
Outcome Measure 30-day and 90-day mortality | From enrollment to 90-day
  Change in 30-day and 90-day mortality (from admission to the ICU until reaching the ninetieth postoperative day)

CONTACTS AND LOCATIONS:
Overall Officials: Jaromir Vajter, Dr., MD, Principal Investigator — University Hospital in Motol
Locations (1):
- University Hospital in Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
No analyzed data are available online. They can be provided after agreement with the principal investigator in case of interest.